CLINICAL TRIAL: NCT07128537
Title: Effectiveness of Oropharyngeal Suctioning in Preventing Ventilator-Associated Pneumonia: A Randomized Controlled Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Hafiz Abdul Wajid, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Health science
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Ventilation Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial (RCT) designed to evaluate the effectiveness of scheduled oropharyngeal suctioning every 4 hours in reducing the incidence of early-onset ventilator-associated pneumonia (VAP) in mechanically ventilated ICU patients. An RCT is the gold standard in clinical research as it helps establish cause-and-effect relationships between an intervention and an outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Oral Care (Twice-Daily Brushing) (Active Comparator): Participants in this group will receive standard oral care as part of ICU routine practice. This includes brushing of teeth, gums, and tongue twice a day to clear accumulated secretions and reduce bacterial growth. Additionally, on-demand suctioning will be performed if clinically indicated (e.g., when visible secretions or discomfort are observed). The control group will not receive the scheduled 4-hourly suctioning intervention, serving as a comparison to evaluate the effectiveness of regular suctioning in preventing VAP.
  Interventions: Procedure: Standard Oral Care (Twice-Daily Brushing)
- Participants in this group will receive scheduled oropharyngeal suctioning every 4 hours, in additio (Experimental): Participants in this group will receive scheduled oropharyngeal suctioning every 4 hours, in addition to routine oral care (twice-daily brushing of teeth, gums, and tongue). The oropharyngeal suctioning involves the mechanical removal of secretions from the oral cavity and pharynx using a sterile suction catheter to prevent bacterial buildup and aspiration into the lungs. This intervention is intended to reduce the risk of early-onset Ventilator-Associated Pneumonia (VAP) by continuously clearing harmful secretions from the airway.
  Interventions: Procedure: Scheduled Oropharyngeal Suctioning Every 4 Hours

INTERVENTIONS:
Procedure: Scheduled Oropharyngeal Suctioning Every 4 Hours — The intervention in this study involves scheduled oropharyngeal suctioning every 4 hours, which distinguishes it from other oral care protocols used in clinical practice. In this arm, patients will receive systematic suctioning of the oropharyngeal area using a sterile suction catheter every 4 hours throughout their ICU stay, starting from the first day of mechanical ventilation. This frequent suctioning is designed to remove accumulated secretions that can harbor bacteria, reducing the risk of aspiration into the lungs, which is a major cause of early-onset Ventilator-Associated Pneumonia (VAP).
  This intervention is not based on clinical need or visible signs of discomfort (as with traditional on-demand suctioning). Instead, it follows a standardized protocol of proactive, scheduled suctioning. The procedure will be performed by trained ICU staff and will involve suctioning for 10-15 seconds per session, ensuring adequate removal of secretions while minimizing patient discomfort. In
  Arms: Participants in this group will receive scheduled oropharyngeal suctioning every 4 hours, in additio
Procedure: Standard Oral Care (Twice-Daily Brushing) — Participants in this group will receive standard oral care as part of ICU routine practice. This includes brushing of teeth, gums, and tongue twice a day to clear accumulated secretions and reduce bacterial growth. Additionally, on-demand suctioning will be performed if clinically indicated (e.g., when visible secretions or discomfort are observed). The control group will not receive the scheduled 4-hourly suctioning intervention, serving as a comparison to evaluate the effectiveness of regular suctioning in preventing VAP.
  Arms: Standard Oral Care (Twice-Daily Brushing)

SUMMARY:
Ventilator-Associated Pneumonia (VAP) is a serious infection that affects patients who are on mechanical ventilation in intensive care units (ICUs). It can increase the risk of death, prolong hospital stays, and lead to higher healthcare costs. This study is designed to evaluate the effectiveness of scheduled oropharyngeal suctioning (removal of secretions from the mouth and throat) every 4 hours in preventing early-onset VAP in ICU patients who require mechanical ventilation for more than 48 hours.

The study will compare two groups of ICU patients: one group will receive scheduled oropharyngeal suctioning every 4 hours in addition to standard oral care, while the other group will receive only standard oral care. The main goal of the study is to determine whether regular suctioning reduces the incidence of VAP, improves patient recovery, and shortens the duration of mechanical ventilation.

This research will help clarify whether adding scheduled suctioning to standard care can prevent VAP and improve clinical outcomes for critically ill patients, potentially leading to better practices in ICU care.

DETAILED DESCRIPTION:
Ventilator-Associated Pneumonia (VAP) is a major healthcare concern in intensive care units (ICUs), affecting patients who require mechanical ventilation. VAP typically develops more than 48 hours after intubation and is caused by the aspiration of contaminated oropharyngeal secretions into the lungs. This infection is associated with increased morbidity, prolonged ICU stays, and higher mortality rates. The incidence of early-onset VAP (developing within the first 4-5 days of ventilation) is particularly concerning due to its association with more virulent pathogens and higher mortality rates. Despite the implementation of preventive measures, early-onset VAP continues to be a significant clinical challenge, necessitating the exploration of more effective interventions.

The primary aim of this study is to assess the effectiveness of scheduled oropharyngeal suctioning every 4 hours in preventing early-onset VAP in mechanically ventilated ICU patients. Oropharyngeal suctioning, which involves the mechanical removal of secretions from the mouth and throat, is a standard procedure in many ICUs to maintain airway patency. However, its role in preventing VAP, especially when performed at fixed intervals, has not been conclusively established. While previous studies have suggested that oropharyngeal suctioning may reduce VAP risk, the optimal frequency and protocol remain unclear.

This study will be conducted as a randomized controlled trial (RCT) at the Institute of Nursing, University of Health Sciences, Lahore, in collaboration with Jinnah Hospital, Lahore. The study will include 100 ICU patients who are expected to be mechanically ventilated for more than 48 hours. The patients will be randomly assigned to two groups:

Intervention Group: Scheduled oropharyngeal suctioning every 4 hours, in addition to routine oral care.

Control Group: Standard oral care, including twice-daily brushing of teeth, gums, and tongue, and on-demand suctioning based on clinical indications.

The study's primary outcome will be the incidence of early-onset VAP, diagnosed using the Modified Clinical Pulmonary Infection Score (MCPIS), a tool widely used in ICUs to diagnose VAP based on clinical symptoms, microbiological findings, and radiographic evidence. Secondary outcomes will include the duration of mechanical ventilation, ICU length of stay, and patient mortality rates.

The study will also assess the effect of the intervention on various factors, including the rate of microbial colonization in the oropharyngeal area, the impact on bacterial load, and the overall health outcomes of ICU patients. By systematically evaluating the role of scheduled oropharyngeal suctioning, the study aims to provide valuable insights into its potential benefits as part of a broader VAP prevention strategy.

The data collection process will be divided into two phases:

Phase 1 (Day 1): Collection of demographic data, baseline MCPIS score, and other clinical variables.

Phase 2 (Day 5): Follow-up to assess the presence or absence of VAP, the length of ICU stay, the duration of mechanical ventilation, and patient mortality.

Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 24. Descriptive statistics will be used to summarize the data, and chi-square or Fisher's Exact Test will be used to compare the incidence of VAP between the two groups. The duration of mechanical ventilation and ICU stay will be analyzed using t-tests or Mann-Whitney U tests, depending on data distribution. A p-value of ≤ 0.05 will be considered statistically significant.

The study will also explore whether the frequency of oropharyngeal suctioning (every 4 hours vs. as needed) is associated with improvements in other clinical outcomes, including reductions in the duration of mechanical ventilation and the length of ICU stay, which would further demonstrate the potential benefits of this intervention in ICU settings.

In addition to its clinical impact, this study aims to contribute to the development of standardized, evidence-based guidelines for oropharyngeal suctioning in ICUs worldwide, potentially leading to improved VAP prevention protocols. If the findings suggest that scheduled oropharyngeal suctioning is effective in preventing VAP, the results could inform clinical practice and guide the development of best practices for oral care in critically ill patients.

The results of this study are expected to have a significant impact on ICU practices, improving patient safety, reducing the incidence of VAP, and lowering healthcare costs associated with VAP-related complications. Moreover, the study could serve as a foundation for future research into oral care interventions and VAP prevention strategies in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients aged 18-75 years.
* Patients expected to require invasive mechanical ventilation for more than 48 hours.
* Modified Clinical Pulmonary Infection Score (MCPIS) ≤ 5 on Day 1, indicating no or minimal signs of infection.
* Ability to comply with the study protocol, including informed consent from patient attendants.

Exclusion Criteria:

* Patients with chronic respiratory diseases (e.g., COPD, asthma).
* Immunocompromised patients (e.g., those with cancer, organ transplant recipients, or on immunosuppressive therapy).
* Patients with ongoing sepsis or severe infections at the time of enrollment.
* Patients who have been on mechanical ventilation for more than 48 hours at the time of ICU admission.
* Pregnant patients or those unable to comply with the study protocol.
* Patients with dental prosthetics or dentures, as these may interfere with the suctioning process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
incidence of early-onset Ventilator-Associated Pneumonia (VAP) in mechanically ventilated ICU patients. | The primary outcome measure, incidence of early-onset VAP, will be assessed from Day 1 to Day 5 of mechanical ventilation in the ICU, specifically during the period of scheduled oropharyngeal suctioning intervention.
  VAP will be diagnosed using the Modified Clinical Pulmonary Infection Score (MCPIS), which evaluates clinical indicators such as body temperature, pulmonary secretions, white blood cell count, the PaO2/FiO2 ratio, and chest radiography findings. A score of ≥6 on the MCPIS indicates the presence of VAP. This primary outcome will help determine whether the intervention (scheduled oropharyngeal suctioning every 4 hours) significantly reduces the incidence of VAP compared to standard oral care practices in ICU patients.

IPD SHARING:
Plan to Share IPD: Undecided